CLINICAL TRIAL: NCT06891183
Title: Percutaneous Thermal Ablation in Treatment of Lung Cancer
Brief Title: Percutaneous Thermal Ablation in Lung Tumors
Acronym: Radiofrequency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman mohamed farid abdelrahman ali, Resident, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Radiofrequency ablation
Record Dates: First submitted 2024-09-12; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Thermal ablation of lung tumors
  Interventions: Radiation: Percutaneous thermal ablation of lung tumors

INTERVENTIONS:
Radiation: Percutaneous thermal ablation of lung tumors — Percutaneous radiofrequency ablation

SUMMARY:
Lung cancer has a high incidence globally, with Egypt having it as the third most common and most lethal cancer, affecting 16.9% of males and 3.8% of females. While surgery is the preferred treatment for stage 1 non-small cell lung cancer due to positive outcomes, it carries significant risks due to patient comorbidities. Non-invasive treatments like radio frequency ablation (RFA) and microwave ablation (MWA) are alternatives for those unable to undergo surgery. These techniques use energy to destroy tumor tissue with minimal invasiveness and can be guided by computed tomography to ensure accurate ablation.

DETAILED DESCRIPTION:
The incidence of lung cancer is one of the highest in the world. In Egypt lung cancer is the third common cancer and the most lethal malignancy in egypt . Where it is responsible for 16.9% and 3.8% of all cancers in males and females respectively.

Surgery is universally accepted as the best choice of therapy in stage 1 non small lung cancer , this is based on favourable outcomes observed in patients who have been surgically treated. However surgery is often high risk procedure because of several comorbidities affecting this cohort of patients.

Therefore non invasive local treatment that makes it possible to avoid resection of functioning parenchyma or prolonged general anaethesia representa key point in management of patients who are not eligible for surgery.

The ablative technologies utilize several sources of energy and different devices to damage targeted tissue using either radio frequency ablation (RFA) or microwave ablation (MWA) which are mini-invasive procedures as they deliver energy to tumour through single or multiple percutaneous needles.

The goal of TA is to induce targeted tissue damage by heating cells to +60 celsius to obtain a complete necrosis of tumour and surrounding tissue, TA may be performed under either conscious sedation or general anaethesia to avoid pain caused by needle insertion and tissue heating.

Computed tomography is today only accurate image guidance method for lung TA, CT guarantees a direct post-procedure .evaluation of ablation, and ground glass opacity is an indicator of extent of ablation achieved to tumour

ELIGIBILITY:
Inclusion Criteria:

* lung cancer smaller than 5 cm
* metastasis to the lung
* patients with lung cancer and multiple comorbidities who are unfit for surgery

Exclusion Criteria:

* lung cancer larger than 5 cm
* lung cancer stage II or more
* patients who cannot tolerate CT guided needle placement for thermal ablation of lung tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy and success | 1 year
  Determination of tumor size in cm after thermal ablation in treatment of patients who are unfit for surgery or have tumors smaller than 5 cm or metastasis to the lung

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahman F Ali, Principal Investigator — Assiut University
Locations (1):
- Faculty of medicine, Asyut, Egypt